CLINICAL TRIAL: NCT03216889
Title: Cognitive Behavioral Therapy for Insomnia to Address Insomnia Symptoms in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00140418
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Insomnia
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Multiple Sclerosis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Experimental): 6 weeks of CBT-I.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Control (Active Comparator): 6 weeks of stretching and thinking games.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Involves attending 1 hour long sessions weekly for 6 weeks. Sessions will be one-on-one or in a group.
  Arms: Cognitive Behavioral Therapy for Insomnia (CBT-I)
Behavioral: Control — Involves attending 1 hour long sessions weekly for 6 weeks. Sessions will involve stretching and thinking games.
  Arms: Control

SUMMARY:
The purpose of this study is to learn if cognitive behavioral therapy for insomnia (CBT-I) will improve sleep quality, fatigue, and quality of life in individuals with multiple sclerosis (MS) with symptoms of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by physician
* Report of difficulty falling asleep, maintaining sleep, or waking up too early at least 3 nights/week for the past 6 months,
* ≥10 on Insomnia Severity Index
* English speaking
* Core at least 24 on the Mini-Mental State Exam (MMSE) to indicate reduced risk of dementia

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea or restless leg syndrome)
* >4 on STOP BANG indicating high risk of sleep apnea
* Increased risk of restless leg syndrome on Restless Legs Syndrome (RLS) Diagnosis Index
* Nervous system disorder other than MS
* Relapse and/or corticosteroid use in past 8 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from Baseline to Week 7
  The ISI consists of 7 questions, each rated on a 0-4 scale. The range of scores on the ISI is 0-28, with a score of ≥ 10 suggesting clinical insomnia. The lower the score the less severe insomnia.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline to Week 7
  The PSQI consists of 9 items within 7 sleep categories. The 7 sleep category scores are summed to form a single global score ranging from 0-21. A global score of >5 reflects poor sleep quality.
Modified Fatigue Impact Scale (MFIS) | Change from Baseline to Week 7
  The MFIS assesses the impact of fatigue on daily activities for the month prior. The MFIS consists of 21 items with 3 subscales: physical, cognitive, and psychosocial. The score on the 21 items are scored with a range of 0-84 with a higher score indicating a greater impact of fatigue.
Fatigue Severity Scale (FSS) | Change from Baseline to Week 7
  The FSS assesses the impact of fatigue on activities for the week prior and consists of 9 questions. The mean of the 9 scores is calculated with a range of 0-7.
Multiple Sclerosis Impact Scale (MSIS) | Change from Baseline to Week 7
  Quality of life will be assessed using the Multiple Sclerosis Impact Scale (MSIS-29). MSIS-29 is total of 29 items scale, with subscales of physical (20 items) and psychological (9 items). Responses computed in a range from 0-100, and higher scores indicating a worse quality of life due to physical and physiological impacts of MS.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Siengsukon, PT, PhD, Study Chair — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States